CLINICAL TRIAL: NCT01743976
Title: Donepezil Compared to Placebo in Patients With Chronic Neuropathic Pain
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Failure to recruit subjects
Sponsor: Wake Forest University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00022107; R01NS057594 (NIH)
Record Dates: First submitted 2012-11-20; First posted 2012-12-06 (Estimated); Results first posted 2020-11-18 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2020-10

CONDITIONS: Neuropathic Pain
Keywords: neuropathic pain; diabetic neuropathy; neuropathic pain after back surgery
MeSH Terms: conditions — Neuralgia; Diabetic Neuropathies | interventions — Donepezil; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Donepezil (Experimental): donepezil 5 mg every day
  Interventions: Drug: Donepezil
- Placebo (Placebo Comparator): Placebo (sugar pill) every day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Donepezil — donepezil 5 mg once daily for 6 weeks
  Other Names: Aricept
  Arms: Donepezil
Drug: Placebo — placebo or sugar pill will be taken once daily for 6 weeks
  Other Names: sugar pill
  Arms: Placebo

SUMMARY:
Based on laboratory studies, donepezil will improve pain relief more than placebo in patients with chronic neuropathic pain who are currently taking gabapentin or pregabalin.

DETAILED DESCRIPTION:
Investigators are currently examining in the laboratory the mechanisms which lead to sprouting of noradrenergic fibers in the spinal cord in models of chronic pain as well as the mechanisms that lead to a novel noradrenergic - cholinergic circuit in the spinal cord. In addition to examining the circumstances which generate this increased capacity for analgesia and the mechanisms by which they occur, investigators will test in this protocol whether approved and experimental treatments for neuropathic pain exploit this increased capacity.

This study is in patients with neuropathic pain taking gabapentin or pregabalin, and will test the clinical relevance of these preclinical data by comparing placebo to the cholinesterase inhibitor. Investigators focus not only on mechanistic hypotheses in the laboratory studies, but also on practical applications, using clinically approved drugs, including gabapentin and pregabalin to activate noradrenergic activity and donepezil (Aricept®), approved for the treatment of Alzheimer's dementia, but not previously tested to treat neuropathic pain, to inhibit cholinesterase. Each of these drugs may act by mechanisms in addition to those involved in descending noradrenergic inhibition, but investigators hypothesize that the therapeutic strength of their combination relies heavily on this cascade engendered by noradrenergic sprouting and altered α2-adrenoceptor function. The proposed studies will provide critical tests of this hypothesis and critical information to guide more effective clinical therapy of neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diabetic neuropathy or failed back syndrome with neuropathic symptoms
* Age 18-80
* Taking a stable dose of gabapentin or pregabalin

Exclusion Criteria:

* Pregnant women or women of child-bearing potential not willing to practice a reliable form of birth control
* Allergy to donepezil or other piperidine derivatives (including fentanyl, alfentanil, sulfentanil, remifentanyl, demerol, tramadol, loperamide, diphenoxylate, betaprodine, alphaprodine, ethopropazine, anileridine, piminodine, 1-methyl-4-phenyl-1,2,3,6-tetrahydropyridine(MPTP),loratadine, fexofenadine
* Unstable medical conditions including cardiac, pulmonary, renal or hepatic diseases that, in the opinion of the investigator, would preclude patients from finishing the trial
* Any person with pending litigation
* A history of major psychosis requiring hospitalization within the last three years
* Non-English speaking, illiterate, unable to comprehend consent
* Lack of contact information
* Uncontrolled narrow-angle glaucoma
* Currently being treatment with thioridazine (Mellaril)
* Patients taking opioids will be excluded if they are taking a dosage that exceeds an equivalent of 30 mg of morphine per day
* Patients taking more than one regular (not rescue) medication for pain
* Patients taking donepezil for dementia
* Patients with a baseline pain score less than 2 (0-10 scale) or greater than 8 (0-10) will be excluded

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2013-10-23 (Actual); Study Completion 2013-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James C Eisenach, M.D., Principal Investigator — Wake Forest University Health Sciences
Locations (2):
- United States (2):
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Donepezil | Placebo
Started | 2 | 3
Completed | 2 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Donepezil | Placebo | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Continuous [Median (Full Range); unit: years] | 44 [38 to 50] | 52 [48 to 69] | 50 [38 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 0 | 2 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 3 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 0 | 1 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: McGill Short Form Pain Questionnaire (SF MPQ) Visual Analog Scale (VAS) Pain Intensity
Description: A greater number is considered a worse outcome. VAS Range (0-10) 0=No Pain 10=The worst pain imaginable.
Time Frame: baseline
Measure: Median (Full Range); unit: units on the scale
Arm/Group | Donepezil | Placebo
Number analyzed (Participants) | 2 | 3
units on the scale | 3.0 [1.3 to 4.7] | 5.0 [4.6 to 5.5]

2. Secondary Outcome: Average From Baseline Profile of Mood States-Short Form (POMS-SF) at 10 Weeks
Description: The questionnaire records total mood disturbance. The scale ranges from 0-100 with a greater number denoting a worse outcome.
Time Frame: baseline, week 8 after baseline, and week 10 after baseline
Measure: Median (Full Range); unit: Total score on POM-S scale
Arm/Group | Donepezil | Placebo
Number analyzed (Participants) | 2 | 3
Total score on POM-S scale
  baseline | 27 [26 to 28] | 53 [23 to 71]
  Week 8 after Baseline | 25 [23 to 27] | 24 [16 to 45]
  Week 10 after Baseline | 33 [27 to 40] | 24 [15 to 38]

3. Secondary Outcome: Number of Days With Rescue Treatment
Description: Questionnaires detailing the amount of rescue pain medications will be completed twice daily.
Time Frame: Days: baseline, week 8 after baseline, and week 10 after baseline
Measure: Median (Full Range); unit: Days
Arm/Group | Donepezil | Placebo
Number analyzed (Participants) | 2 | 3
Days
  Baseline | .5 [0 to 1] | 0 [0 to 2]
  Week 8 after Baseline | 0 [0 to 0] | 0 [0 to 6]
  Week 10 after Baseline | 0 [0 to 0] | 0 [0 to 6]

4. Primary Outcome: McGill Short Form Pain Questionnaire (SF MPQ) Visual Analog Scale (VAS) Pain Intensity
Description: A greater number is considered a worse outcome. VAS Range (0-10) 0=No Pain 10=The worst pain imaginable.
Time Frame: Week 8: last week of study drug treatment
Measure: Median (Full Range); unit: units on the scale
Arm/Group | Donepezil | Placebo
Number analyzed (Participants) | 2 | 3
units on the scale | 0.7 [0.1 to 1.6] | 2.4 [0.1 to 5.4]

5. Primary Outcome: McGill Short Form Pain Questionnaire (SF MPQ) Visual Analog Scale (VAS) Pain Intensity
Description: A greater number is considered a worse outcome. VAS Range (0-10) 0=No Pain 10=The worst pain imaginable.
Time Frame: Week 10: last week of washout
Measure: Median (Full Range); unit: units on the scale
Arm/Group | Donepezil | Placebo
Number analyzed (Participants) | 2 | 3
units on the scale | 0.4 [0.1 to 0.7] | 2.8 [0.1 to 5.2]

ADVERSE EVENTS:
Arm/Group | Donepezil | Placebo
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/3
Other Adverse Events (participants affected / at risk) | 0/2 | 0/3

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2012-11-19): https://cdn.clinicaltrials.gov/large-docs/76/NCT01743976/Prot_SAP_000.pdf
  • Informed Consent Form (2015-09-14): https://cdn.clinicaltrials.gov/large-docs/76/NCT01743976/ICF_001.pdf